CLINICAL TRIAL: NCT06016270
Title: A Phase Ib/II Study of hSTC810 in Combination With Paclitaxel in Relapsed or Refractory Extensive Stage Small Cell Lung Cancer
Brief Title: A Study of hSTC810 in Combination With Paclitaxel in Relapsed or Refractory Extensive Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company strategy
Sponsor: STCube, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STCUBE-002
Record Dates: First submitted 2023-08-17; First posted 2023-08-29 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2023-08

CONDITIONS: Extensive Stage Small Cell Lung Cancer
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- hSTC810 400 mg + Paclitaxel (Experimental): hSTC810 400 mg will be administered with a standard dose of paclitaxel
  Interventions: Drug: hSTC810 400 mg + Paclitaxel
- hSTC810 800 mg + Paclitaxel (Experimental): hSTC810 800 mg will be administered with a standard dose of paclitaxel
  Interventions: Drug: hSTC810 800 mg + Paclitaxel

INTERVENTIONS:
Drug: hSTC810 400 mg + Paclitaxel — hSTC810 400 mg and paclitaxel 175 mg/m2 will be administered as an intravenous (IV) infusion
  Paclitaxel: 175 mg/m2 will be administered as an IV infusion
  Arms: hSTC810 400 mg + Paclitaxel
Drug: hSTC810 800 mg + Paclitaxel — hSTC810 800 mg and paclitaxel 175 mg/m2 will be administered as an IV infusion
  Arms: hSTC810 800 mg + Paclitaxel

SUMMARY:
The purpose of this clinical study is to assess the safety and efficacy of hSTC810 and paclitaxel combination therapy in patients with relapsed or refractory extensive stage small cell lung cancer.

DETAILED DESCRIPTION:
The study will be conducted in 2 parts. Phase Ib will evaluate the safety of the combination of hSTC810 with a standard dose of paclitaxel using a 3+3 dose escalation design. Phase II will evaluate the efficacy of hSTC810 + paclitaxel combination therapy using a Simon 2-stage method.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign an informed consent form
* Male or female ≥ 18 years of age
* Histologically or cytologically confirmed SCLC
* R/R ES-SCLC on or after platinum-based chemotherapy for SCLC with documented disease progression
* At least 1 measurable lesion as defined by RECIST 1.1
* Eastern Cooperative Oncology Group Performance Score (ECOG PS) of 0 or 1
* Life expectancy of at least 3 months
* Adequate organ function as described in the protocol
* For female or male patients with reproductive potential: Agree to use contraception throughout the study and at least 5 months after the last dose.

Exclusion Criteria:

* Known active leptomeningeal disease (carcinomatous meningitis)
* Known active and uncontrolled central nervous system (CNS) metastases
* Treatment with immunotherapy, chemotherapy, targeted small molecule therapy, or any other investigational agent < 14 days prior to initiation of study treatment
* Treatment with radiation therapy < 14 days prior to initiation of study treatment
* Major surgery < 21 days prior to initiation of study treatment
* Received live vaccine < 30 days prior to initiation of study treatment, including intranasal influenza vaccine
* History of another primary malignancy with protocol-defined exceptions
* Active or history of autoimmune disease requiring systemic treatment
* Receiving high doses of steroids or other immunosuppressive medications
* Active hepatitis B or C infection
* Active or history of non-infectious pneumonitis requiring treatment with steroids
* Active uncontrolled viral, fungal, or bacterial infection including tuberculosis
* Pregnant or breastfeeding female patients
* History of severe hypersensitivity reaction to a monoclonal antibody treatment
* History of severe hypersensitivity reaction or ≥ Grade 3 adverse event (AE) to paclitaxel treatment
* History of cerebral vascular event, unstable angina, myocardial infarction, or cardiac symptoms within 6 months prior to screening
* QT Corrected for Fridericia's method (QTcF) > 470 ms at screening
* Lack of resolution of any toxicity to max Grade 1 (except alopecia)
* Active or history of any condition, therapy, or lab abnormality that may interfere with the patient participation for the full duration of the study
* Known psychiatric or substance use disorder
* Positive Coronavirus disease 2019 (COVID-19) test at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 3 months
  Percentage of patients with confirmed Confirmed Response (CR) or Partial Response (PR) as defined by RECIST 1.1 at 3 months
Progression Free Survival (PFS) rate | 6 months
  Proportion of patients without documented progression of disease and alive at 6 months

SECONDARY OUTCOMES:
Safety and tolerability | Up to 4 years
  Incidence, causality, and nature of Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Overall Response Rate (ORR) | Up to 4 years
  Investigator assessed ORR defined by RECIST 1.1
Duration of Response (DoR) | Up to 4 years
  Time from the date of first documented CR or PR until the date of documented progression or death
Progression Free Survival (PFS) | Up to 4 years
  Time from first dose until the date of objective disease progression or death
Clinical Benefit Rate (CBR) | Up to 4 years
  Percentage of evaluable patients with CR, PR, or Stable Disease (SD) lasting ≥ 24 weeks
Overall Survival (OS) | Up to 4 years
  Time from first dose of study drug until the date of death
Overall Survival (OS) rate | 12 months
  Proportion of patients alive at 12 months after the first dose of study drug
Maximum plasma concentration (Cmax) | Up to 21 days
  Maximum plasma concentration of hSTC810 to evaluate PK parameters
Area under the concentration-time curve from 0 to 21 days (AUC0-21) | Up to 21 days
  AUC from 0 to 21 days to evaluate PK parameters
Area under the concentration-time curve extrapolated from 0 to infinity (AUCo-inf) | Up to 21 days
  AUC from time 0 to infinity to evaluate total drug exposure over time
Incidence of anti-drug antibodies (ADA) | Up to 4 years
  Number and percentage of patients with positive ADAs

CONTACTS AND LOCATIONS:
Locations (8):
- United States (2):
  - Tisch Cancer Institute at Mount Sinai, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
- South Korea (6):
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No